CLINICAL TRIAL: NCT01070862
Title: Multiple Myeloma Treatment With Thalidomide. Three Randomized Studies on Thalidomide as Induction Treatment Before Autotransplant (MY-TAG) or With a Conventional Chemotherapy (MY-DECT) and as Consolidation/Maintenance at Plateau Phase (MY-PLAT).
Brief Title: Multiple Myeloma Treated With Thalidomide Before Autotransplant or With Conventional Chemotherapy and as Consolidation/Maintenance Treatment in Young and Elderly Patients : 3 Randomized Studies.
Acronym: MAG 2002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Laphal (Unknown)
Responsible Party: Margaret MACRO, MD, University hospital, Caen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 020879
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Multiple Myeloma de Novo Treatment
Keywords: multiple myeloma, treatment, first line
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Dexamethasone; Vincristine; Doxorubicin; Melphalan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- thalidomide + dexamethasone (Experimental): Thalidomide 200 mg/d at bedtime + Dexamethasone 40 mg/d oral D1-D4 and D15-D18 for 2 first cycles, D1-D4 for the 3d cycle
  Interventions: Drug: Thalidomide, Dexamethasone
- Vincristin, Adriamycin, Dexamethasone (Active Comparator)
  Interventions: Drug: Vincristin , Adriamycin, Dexamethasone = VAD
- thalidomide, melphalan, endoxan, dexamethasone (Experimental)
  Interventions: Drug: Thalidomide, melphalan, endoxan, dexamethasone (MCDex-Thal)
- melphalan, endoxan, dexamethasone (MCDex) (Active Comparator)
  Interventions: Drug: melphalan, endoxan, dexamethasone (MCDex)
- Thalidomide, Dexamethasone (Experimental)
  Interventions: Drug: Thalidomide, Dexamethasone
- watch and wait (No Intervention)

INTERVENTIONS:
Drug: Thalidomide, Dexamethasone — Thalidomide 200 mg/d for 3 months, Dexamethasone 40 mg/d D1-D4 and D14-D17 for 28d-3 cycles
  Arms: thalidomide + dexamethasone
Drug: Vincristin , Adriamycin, Dexamethasone = VAD — Vincristin 0.4 mg/d continUous IV infusion D1-D4, Adriamycin 9 mg/m2 continuous IV infusion D1-D4, Dexamethasone 40 mg/d oral D1-D4 and D15-D18 for 2 first cycles, D1-D4 for the 3d cycle
  Arms: Vincristin, Adriamycin, Dexamethasone
Drug: Thalidomide, melphalan, endoxan, dexamethasone (MCDex-Thal) — Thalidomide : 200 mg/d at bedtime for 3 months , melphalan: 6 mg/m2 oral D1-D4, endoxan 600 mg/m2 IV D1, dexamethasone 40 mg/d oral D1-D4 for 28-d 4 cycles
  Arms: thalidomide, melphalan, endoxan, dexamethasone
Drug: melphalan, endoxan, dexamethasone (MCDex) — melphalan: 6 mg/m2 oral D1-D4, endoxan 600 mg/m2 IV D1, dexamethasone 40 mg/d oral D1-D4 for 28-d 4 cycles
  Arms: melphalan, endoxan, dexamethasone (MCDex)
Drug: Thalidomide, Dexamethasone — Thalidomide 200 mg/d on every other 3 months Dexamethasone 40 mg/d D1-D4, D30-D34,D60-D64, D90-D94
  Arms: Thalidomide, Dexamethasone

SUMMARY:
The aim of the study was to evaluate efficacy and tolerability of Thalidomide in first-line treatment of multiple myeloma as induction treatment in young patients, with Dexamethasone before autotransplant, and in elderly patients in combination with conventional chemotherapy and as consolidation/maintenance therapy in young and elderly patients at plateau-phase.

DETAILED DESCRIPTION:
MY-TAG : Thalidomide as induction treatment before high dose therapy, in young patients MY-DECT : Thalidomide as induction treatment with conventional chemotherapy, in elderly patients MY-PLAT : Thalidomide and Dexamethasone at plateau-phase, after high dose therapy or conventional chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* for MY-TAG(auto-transplant): age 18-65, multiple myeloma Salmon-Durie stage II, stage III and symptomatic stage I (lytic bone lesion or a 25 % increase of monoclonal protein)
* for MY-DECT (conventional chemotherapy) : qge 66-80, multiple myeloma Salmon-Durie stage II, stage III and symptomatic stage I (lytic bone lesion or a 25 % increase of monoclonal protein)
* for MY-PLAT (maintenance at plateau-phase): patients treated in MY-TAG or MY-DECt with at least a minimal response (25 % decrease of M protein)3-6 months after autotransplant or last chemotherapy

Exclusion Criteria:

* for MY-TAG : age 66 or more, smoldering stage I multiple myeloma, previous therapy, plasma cell leukemia,creatinine > 300 micromol/L, liver failure, anthracycline contra-indicated, thalidomide contra-indicated, corticosteroid contra-indicated
* for MY-DECT : age < 66 or > 80, smoldering stage I multiple myeloma, previous therapy, plasma cell leukemia,creatinine > 300 micromol/L, liver failure, thalidomide contra-indicated, corticosteroid contra-indicated
* for MY-PLAT : no response or progressive disease, randomization > 6 m since autotransplant or last chemotherapy, creatinine > 300 micromol/L, liver failure, thalidomide contra-indicated, corticosteroid contra-indicated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-05; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
very good partial response rate (monclonal protein decrease of 90 % or more)at the end induction phase (MY-TAG and MY-DECT), progression free survival during consolidation/maintenance treatment (MY-PLAT) | before autotransplant (MY-TAG), after 4 cycles (MY-DECT), every 6 months (MY-PLAT)

SECONDARY OUTCOMES:
partial response rate (> or = 50%), PFS and OS since diagnosis, safety thalidomide + chemotherapy

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU CAEN Dept of Hematology, Caen
  - CHU Henri Mondor, Créteil
  - CHU Saint Louis Dept of Hematology, Paris